CLINICAL TRIAL: NCT00029848
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose, Multicenter Study of Weight-Reducing Effect and Safety in Obese Patients With Type 2 Diabetes
Brief Title: Obese Patients With Type 2 Diabetes
Acronym: RIO-Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4736
Record Dates: First submitted 2002-01-23; First posted 2002-01-24 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Obesity; Diabetes Mellitus, Non-Insulin-Dependent; Obesity in Diabetes
Keywords: Diabetes; Obesity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rimonabant (SR141716)

SUMMARY:
To assess the effect on weight loss and weight maintenance over a period of one year when prescribed with a hypocaloric diet in obese patients with Type 2 Diabetes

ELIGIBILITY:
* BMI must be greater than 27 and less than 40
* Treated Type 2 Diabetes on single therapy treatment for at least 1 year
* Stable weight (variation of less than 5 kg within 3 months prior to screening visit)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2001-10; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight

SECONDARY OUTCOMES:
Metabolic parameters

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (54):
- United States (44):
  - Innovative Clinical Trials, Birmingham, Alabama
  - Lovelace Scientific Resources, Phoenix, Arizona
  - Advanced Clinicla Therapeutics, LLC, Tucson, Arizona
  - Southern California Prevention and Research Center Inc. (SPARC), Encino, California
  - Anderson Clinical Research, San Bernardino, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - North East Clinical Research, Hamden, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - Jackson Downey, MD, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - DMI Helathcare Group, Largo, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Comprehensive NeuroScience, Inc., Sarasota, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - CSRA Partners in Health, Inc., Augusta, Georgia
  - nTouch Research, Marietta, Georgia
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Physicians Research Group, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Gulf States Clinical Trails, LLC, Kenner, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - Phase III Clinical Research, Fall River, Massachusetts
  - JM Clinical Trials, Inc., Swansea, Massachusetts
  - Twin Cities Clinical Research, Arden Hills, Minnesota
  - Lovelace Scientific Resources, Las Vegas, Nevada
  - Endocrinology and Diabetes Consultants, PC, Dover, New Hampshire
  - Radiant Reseach-Moorestown, Moorestown, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Physician Clinical Research Service, White Plains, New York
  - Center for Nutrition and Preventive Medicine, Charlotte, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - MFP Research, Inc., Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Radiant Research, Portland, Oregon
  - Medical University of South Carolina, Division of Clinical Pharmacology, Charleston, South Carolina
  - Costal Carolina Research Center, Mt. Pleasant, South Carolina
  - TriCities Medical Reseach, Bristol, Tennessee
  - Diabetes $ Glandular Disease Clinic, PA, San Antonio, Texas
  - Endocrine and Diabetes, Ogden, Utah
  - National Clinical Research, Richmond, Virginia
  - Salem Veterans Affairs Medical Center (151), Salem, Virginia
  - The Chase Wellness Center, Inc., Virginia Beach, Virginia
- Sanofi-aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-aventis Administrative Office, Diegem, Belgium
- Sanofi-aventis Administrative Office, Laval, Canada
- Sanofi-aventis Administrative Office, Prague, Czechia
- Sanofi-aventis Administrative Office, Helsinki, Finland
- Sanofi-aventis Administrative Office, Paris, France
- Sanofi-aventis Administrative Office, Berlin, Germany
- Sanofi-aventis Administrative Office, Gouda, Netherlands
- Sanofi-aventis Administrative office, Warsaw, Poland
- Sanofi-aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Scheen AJ, Finer N, Hollander P, Jensen MD, Van Gaal LF; RIO-Diabetes Study Group. Efficacy and tolerability of rimonabant in overweight or obese patients with type 2 diabetes: a randomised controlled study. Lancet. 2006 Nov 11;368(9548):1660-72. doi: 10.1016/S0140-6736(06)69571-8. PMID 17098084